CLINICAL TRIAL: NCT02526472
Title: A Large Prospective Randomized Trial Comparing Trans-abdominal Ultrasound-guided Embryo Transfer (UGET) With a Novel, Modified Trans-vaginal Ultrasound-guided Embryo Transfer Technique (mTVET) Based on Previous Uterine Length Measurement
Brief Title: Transabdominal US-guided (UGET) vs. Modified Transvaginal US-guided (mTVET) Embryo Transfer in Human IVF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Alberto Revelli, Associate Professor, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDR-2-2015
Record Dates: First submitted 2015-08-13; First posted 2015-08-18 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-08

CONDITIONS: Infertility
Keywords: embryo transfer, in vitro fertilization
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- transabdominal US guidance (UGET) (Experimental): ET under transabdominal US guidance (UGET)
  Interventions: Procedure: ET under transabdominal US guidance (UGET)
- TV-US ET guidance (mTVET) (Experimental): ET after transvaginal US uterine measurement (mTVET)
  Interventions: Procedure: ET after transvaginal US uterine measurement (mTVET)

INTERVENTIONS:
Procedure: ET under transabdominal US guidance (UGET) — When UGET was used, a second physician performed trans-abdominal US, and the embryos were discharged when the tip of the catheter was visualized approximately at 1,5 cm from the fundal endometrial surface
  Arms: transabdominal US guidance (UGET)
Procedure: ET after transvaginal US uterine measurement (mTVET) — When mTVET was scheduled, the physician performed a transvaginal US scan just before ET, measured the length of the cervix and of the uterine cavity, and calculated the distance between the internal uterine os and the fundal endometrial surface. Then, ET was performed inserting the inner cannula in order to discharge embryos at a point obtained subtracting 1.5 cm from the total length of the cavity.
  Arms: TV-US ET guidance (mTVET)

SUMMARY:
One thousand, six hundred forty-eight IVF patients undergoing ET with fresh embryos, randomized to receive mTVET (n=828) or UGET (n=820). The transfer in uteri of 1-2 embryos on day 2-3 of culture was performed using a soft catheter either under trans-abdominal US guidance (UGET group) or after measurement of uterine cavity by transvaginal US and calculation of the discharge site (mTVET). Mai outcome measures was the clinical pregnancy rate (CPR), secondary outcomes were the implantation rate (IR), and the patient's discomfort during ET procedure.

DETAILED DESCRIPTION:
All patients undergoing IVF and ending the cycle with the transfer of fresh embryos at investigators' IVF Unit in a 3-years period (n=1824) were proposed to join the study. One hundred forty-six eligible patients refused to sign the consent and were excluded. Overall, 1678 patients accepted to participate in the study and the day of ET were randomized with a 1:1 ratio into two groups using a computer-generated unrestricted randomization: 866 patients were scheduled to undergo UGET, whereas 872 patients were scheduled to receive mTVET. During ET, 90 patients (44 in mTVET group and 46 in UGET group) required to change the catheter for cervical stenosis and consequently were excluded from the analysis. Finally, data of 1648 patients (828 in mTVET group vs. 820 in UGET group) were analyzed.

All cases included in the final analysis were transfers performed on day 2-3 with fresh embryos deriving from autologous IVF. Transfers with frozen embryos and cases in which blastocyst transfer was scheduled were not selected as eligible; donor IVF cycles were not legal in Italy at the time of the study. According to the investigators' usual clinical practice, no mock or trial embryo transfer was performed.

The patient was placed in the lithotomy position, and the cervix was exposed using a speculum. Then, the cervix was gently cleaned using saline solution and the cervical mucus leaking out from the cervical os was removed using a wet gauze.

In order to avoid any bias linked to the operator's experience and skill, all ETs included in the study were performed by three experienced doctors that used the same soft catheter (Sydney®Cook, Melbourne, Australia) loaded by experienced biologists with a constant amount (20 μl) of culture medium. The Sydney catheter was used for all randomized patients, but if cervical stenosis was encountered and ET was difficult, the catheter was changed shifting to a stiffer one. Neither a tenaculum, nor suture points placed on the cervix to pull it were used. All cases with change of the catheter were excluded from the final analysis.

A gentle and slow insertion of the stiffer outer sheath of the catheter was performed, and after inserting the softer inner cannula carrying the embryos, they were gently discharged and the catheter was retracted very slowly. The catheter was immediately and carefully checked under a microscope and if embryos were retained, they were re-harvested to immediately repeat the transfer procedure. These cases were included in the final analysis. The presence of blood inside the cannula was registered. The overall time needed to perform ET (defined as the time elapsed since the loaded catheter was handed by the physician to the time it was returned to the biologist after embryo discharge) was measured and registered.

When UGET was used, a second physician assisted the ET performing trans-abdominal US, and the embryos were discharged when the tip of the catheter was visualized approximately at 1,5 cm from the fundal endometrial surface, which was observed to be the best replacement site according to a previous research by the investigators' group (6).

When mTVET was scheduled, the physician performed a transvaginal US scan using a 6.5 mega-hertz (MHz) transvaginal probe just before ET, visualized the uterus in a sagittal plane, measured the length of the cervix and of the uterine cavity, and calculated the distance between the internal uterine os and the fundal endometrial surface. Then, the probe was taken away from the vagina, a speculum was inserted and ET was performed inserting the inner cannula of the Sydney catheter (that has length markers on it) in order to discharge embryos at a point obtained subtracting 1.5 cm from the total length of the cavity.

Immediately after either UGET or mTVET, the position of the echogenic spot(s) inside the uterus, corresponding to air bubbles loaded with the embryos, was checked by trans-vaginal US, and after waiting approximately 30 seconds its distance (or the distance of a virtual point in the middle of two spots) from the fundal endometrial surface was measured, obtaining the final position of embryo replacement.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing autologous IVF
* ending IVF cycle with the transfer of fresh embryos
* treated at the investigators'r IVF Unit between Jan 2012 to Dec 2014

Exclusion Criteria:

* patients undergoing donor IVF
* ending IVF cycle without embryo transfer
* transferring frozen-thawed embryos
* treated elsewhere

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1648 (Actual)
Dates: Start 2012-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
clinical pregnancy rate per embryo transfer (CPR/ET) | 3 years
implantation rate | 3 weeks (until the pregnancy test is performed)

SECONDARY OUTCOMES:
proportion of patients feeling moderate-to-severe discomfort during ET | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Revelli, Prof., Principal Investigator — Dept. Surgical Sciences, Sant'Anna Hospital, University of Torino, Italy
Locations (1):
- Physiopathology of Reproduction and IVF Unit, S. Anna Hospital, Torino, Italy